CLINICAL TRIAL: NCT05274516
Title: Phase I Clinical Study on the Safety, Tolerability, and Pharmacokinetics of HRS-2261, the Effects of Food on the Pharmacokinetics of HRS-2261, and the Effects of HRS-2261 on CYP3A4 Metabolic Enzymes in Healthy Subjects After Single and Multiple Oral Administration
Brief Title: A Trial of HRS-2261 in Healthy Subjects After Single and Multiple Oral Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-2261-101
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2022-10

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Intervention Model Description: HRS-2261 compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Doses, 6 dose levels (Experimental): HRS-2261 oral tablet Matching placebo to HRS-2261
  Interventions: Drug: HRS-2261 tablet、placebo
- Multiple Ascending Doses, 3 dose levels (Experimental): HRS-2261 oral tablet Matching placebo to HRS-2261
  Interventions: Drug: HRS-2261 tablet、placebo

INTERVENTIONS:
Drug: HRS-2261 tablet、placebo — HRS-2261 oral tablet, oral, single dose. Matching placebo to HRS-2261, oral, single dose.
  Arms: Single Ascending Doses, 6 dose levels
Drug: HRS-2261 tablet、placebo — HRS-2261 oral tablet, oral, BID. Matching placebo to HRS-2261, oral, BID.
  Arms: Multiple Ascending Doses, 3 dose levels

SUMMARY:
This is a first-in-human study that will investigate the safety, tolerability and pharmacokinetics of single and multiple ascending doses of HRS-2261 using a double blind, placebo controlled, randomized study design. The influence of food on the pharmacokinetics of HRS-2261 and the effects of HRS-2261 on CYP3A4 metabolic enzymes will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Age 18 to 55 years (inclusive).
3. Weight of male subjects ≥50 kg, female ≥45kg, body mass index (BMI) 19-26 kg/m2 (inclusive).
4. Medical examination (including physical examination, vital signs, laboratory examination, 12-lead electrocardiogram, abdominal B-ultrasound and chest radiography) normal or abnormal with no clinical significance.

Exclusion Criteria:

1. Any clinically serious diseases such as circulatory, endocrine, nervous, digestive, respiratory, blood, immune, mental and metabolic abnormalities or any other diseases that investigator determines may interfere with the test results.
2. Subjects with severe infection, severe trauma or major surgical operation within 3 months prior to screening; Subjects who plan to undergo surgery during the trial period and within two weeks after the trial.
3. Treated with any drug that inhibits or induces drug metabolism in the liver within 1 month prior to administration.
4. Subjects have any condition or medical condition that affects absorption, metabolism, and/or excretion of the study drug according to the investigator.
5. Subjects enrolled in clinical trials of any drug or medical device within 3 months prior to screening, or within 5 half-lives of the drug before screening.
6. Subjects who had a history of smoking in the previous 3 months (average daily smoking > 5 cigarettes), or who could not stop using any tobacco products during the test period.
7. Subjects who consumed more than 15g of alcohol per day on average (15g of alcohol is equivalent to 450 mL beer, 150 mL wine or about 50mL low-alcohol white wine) or tested positive for alcohol during the 3 months prior to screening, or who could not abstain from alcohol during the test period.
8. Subjects with a history of drug abuse, drug dependence or positive drug screening.
9. Determined by the investigator to be unfit to participate in this clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Number and severity of treatment emergent adverse events (TEAEs) | up to 7 days after the last dose
  Number and severity of TEAEs collected from dosing until follow up 7 days after last dose

SECONDARY OUTCOMES:
Area under the curve (AUC) | up to 7 days after the last dose
  To assess AUC of single and multiple ascending oral doses of HRS-2261
Maximum plasma concentration (Cmax) | up to 7 days after the last dose
  To assess Cmax of single and multiple ascending oral doses of HRS-2261
Area under the curve (AUC) under fed conditions | up to 7 days after the last dose
  To assess AUC of a single oral dose of HRS-2261 under fed conditions
Maximum plasma concentration (Cmax) under fed conditions | up to 7 days after the last dose
  To assess Cmax of a single oral dose of HRS-2261 under fed conditions

CONTACTS AND LOCATIONS:
Locations (1):
- The second hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fan Y, Zhang X, Zhang Q, Zheng L, Zhou R, Sun C, Wang X, Song K, He Z, Wang H, Zhang Q, Hu W. Safety and Pharmacokinetics of HRS-2261, a P2X3 Receptor Antagonist, in Healthy Subjects: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Study. Clin Pharmacokinet. 2024 Mar;63(3):293-302. doi: 10.1007/s40262-023-01330-7. Epub 2024 Jan 10. PMID 38198010